CLINICAL TRIAL: NCT02992886
Title: Multicenter, Phase II Study of Preoperative Chemoradiotherapy With Raltitrexed for Intermediate or Locally Advanced Rectal Cancer in the Fit Elderly
Brief Title: Preoperative Chemoradiotherapy With Raltitrexed for Intermediate or Locally Advanced Rectal Cancer in the Fit Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Jin, M.D., Vice Chair of Radiation Oncology, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-098
Record Dates: First submitted 2016-11-30; First posted 2016-12-14 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Rectal Neoplasms Malignant
Keywords: elderly patients; rectal cancer; preoperative chemoradiotherapy; comprehensive geriatric assessment
MeSH Terms: conditions — Rectal Neoplasms | interventions — raltitrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- preCRT+surgery (Experimental): Treatment including preoperative chemoradiotherapy (preoperative radiation with concurrent chemotherapy) with Raltitrexed followed by surgery. Radiotherapy will be delivered to a planning target volume with a dose of 45-50.4Gy (1.8-2.0Gy daily) using with Intensity-Modulated Radiotherapy or Volumetric-Modulated Arc Therapy technique. During the radiation treatment, concurrent chemotherapy will be delivered (Raltitrexed, intravenous infusion, 3 mg/m2, on d1 and d22). Pelvic surgery is planned 6 weeks after completion of CRT based on the decision of MDT.
  Interventions: Radiation: Preoperative radiation; Drug: Raltitrexed; Procedure: Pelvic surgery

INTERVENTIONS:
Radiation: Preoperative radiation — Radiation treatment before surgery
  Other Names: Preoperative radiotherapy
Drug: Raltitrexed — concurrent chemotherapy
  Other Names: Raltitrexed Injection
Procedure: Pelvic surgery

SUMMARY:
The aim of this multicenter phase II study is to evaluate the response rate, local control, disease-free survival and treatment-related toxicity of preoperative chemoradiation for intermediate or locally advanced rectal cancer in the fit elderly.

DETAILED DESCRIPTION:
The concurrent chemoradiotherapy has become the standard treatment for patients with intermediate or locally advanced rectal cancer. However, the data from prospective trial for elderly patients is still lacking.

The aim of this multicenter phase II study is to evaluate the response rate, local control, disease-free survival and treatment-related toxicity of preoperative chemoradiation with Raltitrexed for intermediate or locally advanced rectal cancer in the fit elderly aged 70 years above.

And all the participants have to be evaluated by comprehensive geriatric assessment (CGA). Clinical stage was evaluated by chest and abdominal computed tomography, endorectal ultrasound, and/or pelvic magnetic resonance imaging.

5 weeks after the preCRT, the multi-disciplinary team decided the following treatment of patients based on imaging evaluation. Surgical resection would be done with a minimum interval of 6 weeks after the last radiation. Acute toxicity was evaluated during and within 2 weeks after CRT. Toxicities were assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0.

Sample size consideration.It has been calculated that 68 patients will need to be included, according to the following assumptions:

Recruitment period of 24 months. Minimum follow-up period of 24 months. We estimated that 51 patients were required to test the hypothesis that the 2-year DFS was equal to or greater than 78% with 80% power and to reject the hypothesis that the 2-year DFS rate was less than 63% at a significance level of 5% (one sided).Taking into account that a 5% percentage of losses, 20% of patients will refuse surgery, 68 patients are expected to be included in the study.

The interim analysis design. An interim safety evaluation will be carried out when 39 patients have finished their preoperative CRT. As the tolerance of elderly patients for nonhematological toxicities (such as diarrhoea) was often more poor than hematological toxicities, we estimated that 39 patients were required to test the hypothesis that the nonhematological G3 or higher acute toxicities rate was equal to or less than 21% ( safety result of patients aged 70 years or older from ACCOR12/PRODIGE 2 phase III trial) with 80% power and to reject the hypothesis that the rate was more than 36% at a significance level of 10% (one sided). If nonhematological G3 or higher acute toxicites is observed in12 or more patients, the H0 hypothesis will be rejected, and the protocal should be re-evaluated.

Biospecimen Retention. Blood, plasma, feces and tissue (optional). Feces were collected before any treatment. Peripheral blood samples of 10-20mL were collected from the patients for CTCs analysis, exploration analysis for frailty and tumor marker before and after preCRT, before and after surgery, and then on each follow up visit, according to our study protocal.

ELIGIBILITY:
* Inclusion Criteria:

  * Rectal adenocarcinoma, clinical stage II/III(T3-4 or N+, AJCC 7th), and fulfils the intermediate or locally advanced risk category standard of ESMO recal cancer clinical practice guidelines 2013.
  * KPS status no less than 70; Charlson comorbidity no more than 2; Fit status evaluated by CGA.
  * Life expectancy more than 6 months.
  * Hemoglobin >= 100g/L, white blood cell >= 3.5*10E9/L, neutrophil >= 1.5*10E9/L, platelet >= 100*10E9/L.
  * Creatin normal, Total bilirubin normal, AST and AST normal, AKP normal.
  * Do not receive surgery ( except palliative colostomy) or chemotherapy or other anti-cancer treatment.
  * No previously pelvic irradiation history.
  * Through MDT discussion, the patient is considered to be candidate for preoperative CRT followed by surgery.
  * Informed consent signed.
* Exclusion Criteria:

  * Other cancer history, except curable non-melanoma skin cancer or cervix in-situ carcinoma.
  * Allergy history to analog of quinazoline folate.
  * Active infection existed.
  * Severe complication, such as acute myocardial infarction in 6 months, uncontrolled diabetes ( Plasma glucose concentrations in any time of a day≥11.1mmol/L）, severe cardiac arrhythmia, etc.
  * Anticipate other clinical trials in four weeks before enrollment.

Min Age: 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-09; Primary Completion 2021-05 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
2-year disease-free survival probability (%) | 2 year
  The probability of staying free from recurrence at 2 year after surgery or clinical complete response of tumor validated on imaging or pathological examination.

SECONDARY OUTCOMES:
5-year overall survival probability | 5 year
  The probability of staying alive at 5 year after surgery or end of CRT (for those who did not receive surgery).
5-year cancer-specific survival probability | 5 year
  The probability of staying free from death caused by cancer at 5 year after surgery or end of CRT (for those who did not receive surgery).
The ratio of patients occured pCR | 2 weeks after surgery
  The ratio of patients occured pathological complete response of tumor.
The ratio of patients occured Grade 3 or higher adverse events. | During chemoradiotherapy and within 180 days after surgery
QOL | Before and after chemoradiotherapy and surgery, and then follow up for 3 years
  The quality of life assessment score by EORTC QLQ-C30 and EORTC QLQ-CR29.

OTHER OUTCOMES:
Exploratory endpoints | 5 years
  To investigate the biomarker from blood or feces (such as circulating tumor cells, circulating tumor DNA) for treatment response and prognosis predicting. To investigate the CGA elements, and willingness evaluation to surgery for predicting the adherence, tolerence and prognosis of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Jin, MD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Department of Radiation Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papamichael D, Audisio RA, Glimelius B, de Gramont A, Glynne-Jones R, Haller D, Kohne CH, Rostoft S, Lemmens V, Mitry E, Rutten H, Sargent D, Sastre J, Seymour M, Starling N, Van Cutsem E, Aapro M. Treatment of colorectal cancer in older patients: International Society of Geriatric Oncology (SIOG) consensus recommendations 2013. Ann Oncol. 2015 Mar;26(3):463-76. doi: 10.1093/annonc/mdu253. Epub 2014 Jul 11. PMID 25015334
- [Background] Li M, Gu J. Changing patterns of colorectal cancer in China over a period of 20 years. World J Gastroenterol. 2005 Aug 14;11(30):4685-8. doi: 10.3748/wjg.v11.i30.4685. PMID 16094710
- [Background] Fiorica F, Cartei F, Licata A, Enea M, Ursino S, Colosimo C, Camma C. Can chemotherapy concomitantly delivered with radiotherapy improve survival of patients with resectable rectal cancer? A meta-analysis of literature data. Cancer Treat Rev. 2010 Nov;36(7):539-49. doi: 10.1016/j.ctrv.2010.03.002. Epub 2010 Mar 23. PMID 20334979
- [Background] Bosset JF, Collette L, Calais G, Mineur L, Maingon P, Radosevic-Jelic L, Daban A, Bardet E, Beny A, Ollier JC; EORTC Radiotherapy Group Trial 22921. Chemotherapy with preoperative radiotherapy in rectal cancer. N Engl J Med. 2006 Sep 14;355(11):1114-23. doi: 10.1056/NEJMoa060829. PMID 16971718
- [Background] Gerard JP, Conroy T, Bonnetain F, Bouche O, Chapet O, Closon-Dejardin MT, Untereiner M, Leduc B, Francois E, Maurel J, Seitz JF, Buecher B, Mackiewicz R, Ducreux M, Bedenne L. Preoperative radiotherapy with or without concurrent fluorouracil and leucovorin in T3-4 rectal cancers: results of FFCD 9203. J Clin Oncol. 2006 Oct 1;24(28):4620-5. doi: 10.1200/JCO.2006.06.7629. PMID 17008704
- [Background] Sebag-Montefiore D, Stephens RJ, Steele R, Monson J, Grieve R, Khanna S, Quirke P, Couture J, de Metz C, Myint AS, Bessell E, Griffiths G, Thompson LC, Parmar M. Preoperative radiotherapy versus selective postoperative chemoradiotherapy in patients with rectal cancer (MRC CR07 and NCIC-CTG C016): a multicentre, randomised trial. Lancet. 2009 Mar 7;373(9666):811-20. doi: 10.1016/S0140-6736(09)60484-0. PMID 19269519
- [Background] Teoh S, Muirhead R. Rectal Radiotherapy--Intensity-modulated Radiotherapy Delivery, Delineation and Doses. Clin Oncol (R Coll Radiol). 2016 Feb;28(2):93-102. doi: 10.1016/j.clon.2015.10.012. Epub 2015 Nov 28. PMID 26643092
- [Background] Tang Y, Liu WY, Jin J, Zhang HZ, Yang L, Ren H, Fang H, Wang WH, Song YW, Liu YP, Wang SL, Li YX. Preoperative chemoradiation with capecitabine for rectal cancer in elderly patients: a phase I trial. Int J Colorectal Dis. 2016 Aug;31(8):1547-9. doi: 10.1007/s00384-016-2577-7. Epub 2016 Apr 8. No abstract available. PMID 27059037
- [Background] Thomas RJ, Williams M, Garcia-Vargas J. Lessons learned from raltitrexed--quality assurance, patient education and intensive supportive drugs to optimise tolerability. Clin Oncol (R Coll Radiol). 2003 Aug;15(5):227-32. doi: 10.1016/s0936-6555(03)00092-x. PMID 12924450
- [Background] Cunningham D, Zalcberg J, Maroun J, James R, Clarke S, Maughan TS, Vincent M, Schulz J, Gonzalez Baron M, Facchini T. Efficacy, tolerability and management of raltitrexed (Tomudex) monotherapy in patients with advanced colorectal cancer. a review of phase II/III trials. Eur J Cancer. 2002 Mar;38(4):478-86. doi: 10.1016/s0959-8049(01)00413-0. PMID 11872339
- [Background] Feliu J, Mel JR, Camps C, Escudero P, Aparicio J, Menendez D, Garcia Giron C, Rodriguez MR, Sanchez JJ, Gonzalez Baron M; Oncopaz Cooperative Group Associated Hospitals. Raltitrexed in the treatment of elderly patients with advanced colorectal cancer: an active and low toxicity regimen. Eur J Cancer. 2002 Jun;38(9):1204-11. doi: 10.1016/s0959-8049(02)00005-9. PMID 12044507
- [Background] Valentini V, Doglietto GB, Morganti AG, Turriziani A, Smaniotto D, De Santis M, Ratto C, Sofo L, Cellini N. Preoperative chemoradiation with raltitrexed ('Tomudex') for T2/N+ and T3/N+ rectal cancers: a phase I study. Eur J Cancer. 2001 Nov;37(16):2050-5. doi: 10.1016/s0959-8049(01)00247-7. PMID 11597383
- [Background] Valentini V, Coco C, Minsky BD, Gambacorta MA, Cosimelli M, Bellavita R, Morganti AG, La Torre G, Trodella L, Genovesi D, Portaluri M, Maurizi-Enrici R, Barbera F, Maranzano E, Lupattelli M. Randomized, multicenter, phase IIb study of preoperative chemoradiotherapy in T3 mid-distal rectal cancer: raltitrexed + oxaliplatin + radiotherapy versus cisplatin + 5-fluorouracil + radiotherapy. Int J Radiat Oncol Biol Phys. 2008 Feb 1;70(2):403-12. doi: 10.1016/j.ijrobp.2007.06.025. Epub 2007 Oct 4. PMID 17919844
- [Background] Francois E, Azria D, Gourgou-Bourgade S, Jarlier M, Martel-Laffay I, Hennequin C, Etienne PL, Vendrely V, Seitz JF, Conroy T, Juzyna B, Gerard JP. Results in the elderly with locally advanced rectal cancer from the ACCOR12/PRODIGE 2 phase III trial: tolerance and efficacy. Radiother Oncol. 2014 Jan;110(1):144-9. doi: 10.1016/j.radonc.2013.10.019. Epub 2014 Jan 10. PMID 24418359
- [Background] Glimelius B, Tiret E, Cervantes A, Arnold D; ESMO Guidelines Working Group. Rectal cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2013 Oct;24 Suppl 6:vi81-8. doi: 10.1093/annonc/mdt240. No abstract available. PMID 24078665
- [Derived] Liu WY, Tang Y, Li N, Tang Y, Cheng YJ, Yang L, Fang H, Lu NN, Qi SN, Chen B, Wang SL, Song YW, Liu YP, Li YX, Liu Z, Liang JW, Pei W, Wang XS, Zhang HZ, Wang J, Zhou HT, Jin J. Preoperative chemoradiotherapy in older patients with rectal cancer guided by comprehensive geriatric assessment within a multidisciplinary team-a multicenter phase II trial. BMC Geriatr. 2024 May 21;24(1):442. doi: 10.1186/s12877-024-05046-6. PMID 38773457